CLINICAL TRIAL: NCT02637661
Title: Earlobe Crease as Risk Factors of Acute Myocardial Infarction in Chinese Population
Acronym: ELC-AMI-CHN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Jing Qi (Other)
Collaborators: General Hospital of Shenyang Military Region (Other); Beihua University (Other); Zhejiang Provincial Tongde Hospital (Other); Zhejiang Chinese Medical University (Other Government)
Responsible Party: Sponsor-Investigator, Jing Qi, Principal investigator, Liaoning University of Traditional Chinese Medicine
Organization: Liaoning University of Traditional Chinese Medicine (Other)
Other Study IDs: JQi1
Record Dates: First submitted 2015-11-30; First posted 2015-12-22 (Estimated); Last update posted 2016-01-11 (Estimated); Status verified 2016-01

CONDITIONS: Ear/*Abnormalities; Risk Factor
Keywords: earlobe crease; acute myocardial infarction; risk factor

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Initial AMI: To study the sensitivity, specificity, positive predictive value, and negative predictive value of different earlobe crease as risk factors of AMI
  Interventions: Other: earlobe crease positive; Other: earlobe crease negative
- No coronary heart disease: To study the characteristics of earlobe crease
  Interventions: Other: earlobe crease positive; Other: earlobe crease negative

INTERVENTIONS:
Other: earlobe crease positive
Other: earlobe crease negative

SUMMARY:
The purpose of this study is to explore the earlobe crease as a risk factor of acute myocardial infarction (AMI)in the Chinese population, combined with other risk factors, to predict high risk patients with coronary heart disease.

DETAILED DESCRIPTION:
Primary objectives: Odds ratio and 95% confidence interval of binaural earlobe crease as risk factors of AMI.

Secondary objectives:

1. To study the characteristics of different earlobe creases in different gender of the patients with AMI.
2. To analyze the characteristics of earlobe crease in different age groups.
3. To compare the feature of earlobe crease in acute ST elevation myocardial infarction and non ST elevation myocardial infarction.
4. The sensitivity,specificity,positive likelihood ratio and negative likelihood ratio of binaural earlobe crease as risk factors of AMI.

ELIGIBILITY:
Inclusion Criteria:

1. Initial acute myocardial infarction(AMI).
2. Detection of a rise and/or fall of cardiac biomarker values (preferably cardiac troponin(cTn) with at least one value above the 99th percentile upper reference limit(URL)) and with at least one of the following:

   * Symptoms of ischemia
   * Development of pathologic Q waves in the electrocardiogram (ECG)
   * New or presumed new significant ST-segment-T wave (ST-T) changes or new left bundle branch block (LBBB).
   * Identification of an intracoronary thrombus by angiography or autopsy
   * Imaging evidence of new loss of viable myocardium or a new regional wall motion abnormality.
3. Type 1 (spontaneous myocardial infarction(MI)) in the third universal definition of MI: MI consequent to a pathologic process in the wall of the coronary artery (eg, plaque erosion/rupture, fissuring, or dissection), resulting in intraluminal thrombus.
4. Infarct related artery (IRA) showed that acute thrombus formation, IRA occlusion or stenosis ≥95%、≥90%～95%、≤90%，thrombolysis in myocardial infarction(TIMI) 0-3 flow.
5. Signed informed consent.

Exclusion Criteria:

1. Combined valvular heart disease, cardiomyopathy, blood diseases, skin diseases, rheumatic diseases, ischemic cerebrovascular disease, tumor, etc.
2. Previous myocardial infarction.
3. Previous percutaneous coronary intervention(PCI) and coronary artery bypass graft(CABG).
4. Chronic total occlusion(CTO)lesions.
5. Ear malformation.
6. Ocular diseases.
7. Participating in a clinical study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The case group is Initial acute myocardial infarction(AMI),the control group is no coronary heart disease
Sampling Method: Probability Sample
Enrollment: 236 (Estimated)
Dates: Start 2015-06; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Odds ratio(OR，the ratio of the explosure number and non-explosure in case group/ the ratio of the explosure number and non-explosure in control group) and 95% confidence interval were calculated of binaural earlobe crease≥ 7 scores as risk factors of AMI | 3 years

SECONDARY OUTCOMES:
The score of the ELC in different gender of the patients with AMI. | 3 years
The score of ELC in different age groups. | 3 years
To compare the score of the ELC in acute ST elevation myocardial infarction and non ST elevation myocardial infarction. | 3 years
The sensitivity(true positive/true positive+false negative) and specificity(true negative/true negative+false positive) of binaural earlobe crease≥ 7 scores as risk factors of AMI. | 3 years
Positive likelihood ratio(+LR，sensitivity/1-speccificity)and negative likelihood ratio(-LR，1-sensitivity/specificity)of binaural earlobe crease≥ 7 scores as risk factors of AMI | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Junwen Jiang, Doctor, Principal Investigator — Liaoning University of Traditional Chinese Medecine
Locations (1):
- Jing, Shenyang, Liaoning, China